CLINICAL TRIAL: NCT04076995
Title: INDIGO-2: The Effect of High Water Intake on Glucose Regulation in Low-drinkers
Acronym: INDIGO-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00010276
Record Dates: First submitted 2019-08-27; First posted 2019-09-04 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Dehydration; Diabetes Mellitus, Type 2
Keywords: dehydration; vasopressin; copeptin
MeSH Terms: conditions — Dehydration; Diabetes Mellitus, Type 2; Diabetes Insipidus | interventions — Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Water intake (Experimental): High water intake of 3.0 L/day in males and 2.0 L/day in females
  Interventions: Other: Water Intake
- Low Water Intake (Active Comparator): Low water intake of 0.5 L/day in males and 0.4 L/day
  Interventions: Other: Water Intake

INTERVENTIONS:
Other: Water Intake — Increased water intake during the 11 h protocol

SUMMARY:
Previous studies have indicated increased vasopressin due to hypertonic saline infusion impairs glucose regulation. The current study will examine the effect of low water intake on glucose regulation. No currently published study has investigated the acute effect of low water intake on glucose regulation using continuous glucose monitoring over the course of a full day. The aim of the study is to observe the effect of low water intake on glucose regulation in low drinkers. The study will study the glycemic responses to standardized meals in adults during an 11-hour period in two conditions: a) high water intake and b) low water intake. It is hypothesized that the area under the glucose curve will be greater in the low water intake trial as compared to the high water intake trial

ELIGIBILITY:
Inclusion Criteria:

* healthy sedentary participants
* aged 30-55 years
* body mass 27.5-35.0 kg·m2
* low water intake less than 1.5 L∙day-1 (male) or 1.0 L∙day-1 (female)
* 24 h urine osmolality greater than 800 mmol/kg

Exclusion Criteria:

* diabetes HbA1c >6.5%
* impaired liver or kidney function
* cardiovascular disease
* weight change of more than 3 kg in the past month
* pregnancy
* previous surgery on digestive tract
* exercise >4 h/week

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Area under the curve of Glucose at lunch | 2-hour window starting right before the lunch meal (12:00 pm - 2:00 pm)
Area under the curve of Glucose at Dinner | 2-hour window starting right before dinner (4:00 pm - 6:00 pm)
Area under the curve of Glucose for the entire experiment | 11-hour window starting right before breakfast till 2 hours after dinner (7:00 am - 6:00 pm)
Area under the curve of Copeptin for the entire experiment | 11-hour window starting right before breakfast till 2 hours after dinner (7:00 am - 6:00 pm)
Area under the curve of Glucagon at lunch | 2-hour window starting right before the lunch meal (12:00 pm - 2:00 pm)
Area under the curve of Glucagon at dinner | 2-hour window starting right before dinner (4:00 pm - 6:00 pm)
Urinary glucose excretion | Entire 11-hour protocol 7:00 am - 6:00 pm
Area Under the Curve for Plasma osmolality | the entire 11-hour protocol 7:00 am - 6:00 pm

SECONDARY OUTCOMES:
Area under the curve of Insulin at lunch | 2-hour window starting right before the lunch meal (12:00 pm - 2:00 pm)
Area under the curve of Insulin at dinner | 2-hour window starting right before dinner (4:00 pm - 6:00 pm)
Area under the curve of Glucagon like peptide 1 at dinner | 2-hour window starting right before dinner (4:00 pm - 6:00 pm)
Area under the curve of Glucagon like peptide 1at lunch | 2-hour window starting right before the lunch meal (12:00 pm - 2:00 pm)
Area under the curve of plasma cortisol | the entire 11-hour protocol 7:00 am - 6:00 pm
Area under the curve for Thirst rating | the entire 11-hour protocol 7:00 am - 6:00 pm
  Thirst assessed by Visual analog scale
Mood assessment with a questionnaire | single measurement at baseline before the beginning of breakfast at 7:00 am and 1-hour before dinner meal at 3:00 pm
  Assessed by Profile of mood state questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No